CLINICAL TRIAL: NCT00280553
Title: A Pilot Study of Bupivacaine Infusion in Abdominal Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Margherita CADDEDU (Other)
Collaborators: McMaster University (Other); The Physicians' Services Incorporated Foundation (Other); St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor-Investigator, Margherita CADDEDU, MD, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04-2399
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Laparoscopic Surgical Procedures
Keywords: analgesia; laparoscopic surgical procedures; length of stay
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- patient controlled analgesia (PCA) only (No Intervention)
- PCA and pump with saline infusion for up to five days (Other)
  Interventions: Other: Saline infusion
- PCA and bupivicaine infusion for up to five days (Other)
  Interventions: Drug: bupivicaine

INTERVENTIONS:
Drug: bupivicaine — PCA and bupivicaine infusion for up to five days
  Arms: PCA and bupivicaine infusion for up to five days
Other: Saline infusion — PCA and pump with saline infusion for up to five days
  Arms: PCA and pump with saline infusion for up to five days

SUMMARY:
The incisions used in abdominal surgery can be quite painful, requiring strong pain medications. A new pain pump that trickles small amounts of local freezing into the incision has been developed that helps numb the area so that the patient does not feel the pain for two to five days after surgery.

The main research question is whether use of the pain pump will result in decreased hospital length of stay. The research is important because if the pain pump is found to be effective, it can substantially decrease the length of stay. Areas to be studied include hospital length of stay, patient's comfort post-operatively, and post-operative complications.

DETAILED DESCRIPTION:
Pain in the post-operative period has been a limiting factor delaying recovery following abdominal surgery. Furthermore, it has been associated with several complications including ileus, urinary retention, delay to tolerating oral intake and enteral feeds, thrombo-embolic complications, and respiratory complications such as atelectasis and pneumonia. Diminishing pain in the post-operative period has been a subject of great study and to date the role of epidural analgesia, epidural anesthesia, patient controlled anesthesia and narcotic analgesia has been well documented to assist in controlling pain, decreasing morbidity and accelerating recovery in the post-operative period following colorectal surgery.

Nevertheless, the use of opioid-based analgesic techniques via epidural, nurse or patient controlled delivery systems either oral or parenteral can produce adverse effects such as nausea, vomiting, ileus, delay in tolerance or urinary retention. Concomitant use of non-narcotic based analgesics have failed to obviate the need for narcotic based analgesia. Recently, several companies have developed devices that deliver a constant rate of local anesthetic via a spring loaded device through a multiport catheter inserted into the incision. The effectiveness of these bupivicaine infusion pumps has been demonstrated to diminish post-operative pain following orthopedic, plastic, thoracic and cardiac surgeries but to date their role has not been evaluated in colorectal surgery or abdominal surgery.

The rational of the study is that bupivicaine infusion pumps are being used at St. Joseph's Healthcare for patients undergoing laparoscopic assisted colorectal surgery, and anecdotally, the patients have less pain, need less narcotics and can ambulate and be discharged sooner. This pilot study aims to gather prospective randomized data regarding post-operative length of stay and patient pain scores so that a properly powered randomization study can be undertaken to understand if the bupivicaine infusion system helps decrease length of stay and patient's post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* eligible and consented patients between the ages of 18 and 80
* male and female patients
* scheduled for elective laparoscopic colorectal resection
* anesthetist-assessed to be ASA 1-3

Exclusion Criteria:

* patients with allergies to medications used in study
* non-ambulatory patients
* patients with foreign bodies (ie. Orthopedics prostheses)
* patients requiring colostomies as part of procedure
* patients with enterocutaneous, entero-enteric, enterovaginal, enterovesicular, recto-vaginal, entero-utero fistulas
* pregnant patients
* immuno-compromised patients
* patients with moderate to severe ascites or moderate to severe hepatic insufficiency
* patients unable to speak and comprehend English
* patients requiring emergency colorectal resection
* patients who, for medical reasons assessed by an anesthetist, are deemed deserving of epidural analgesia
* patients with seizure disorders
* patients assessed by an anesthetist to be ASA 4 or 5

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
length of stay postoperative in hospital | end of surgery to discharge

SECONDARY OUTCOMES:
subjective pain of patient | Pre-op and post-op
incidence of in-hospital and post-discharge complications | Post-op days 1, 2, 3, 5 and 14
amount of narcotic and non-narcotic analgesia required | Post-op 1, 2, 3, 5 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Margherita Cadeddu, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University-St. Joseph's Healthcare, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Skinner HB, Shintani EY. Results of a multimodal analgesic trial involving patients with total hip or total knee arthroplasty. Am J Orthop (Belle Mead NJ). 2004 Feb;33(2):85-92; discussion 92. PMID 15005598
- [Background] Carabine UA, Gilliland H, Johnston JR, McGuigan J. Pain relief for thoracotomy. Comparison of morphine requirements using an extrapleural infusion of bupivacaine. Reg Anesth. 1995 Sep-Oct;20(5):412-7. PMID 8519719
- [Background] Baroody M, Tameo MN, Dabb RW. Efficacy of the pain pump catheter in immediate autologous breast reconstruction. Plast Reconstr Surg. 2004 Sep 15;114(4):895-8; discussion 899-900. doi: 10.1097/01.prs.0000133173.71201.3c. PMID 15468395
- [Background] White PF, Rawal S, Latham P, Markowitz S, Issioui T, Chi L, Dellaria S, Shi C, Morse L, Ing C. Use of a continuous local anesthetic infusion for pain management after median sternotomy. Anesthesiology. 2003 Oct;99(4):918-23. doi: 10.1097/00000542-200310000-00026. PMID 14508326
- [Background] Cheong WK, Seow-Choen F, Eu KW, Tang CL, Heah SM. Randomized clinical trial of local bupivacaine perfusion versus parenteral morphine infusion for pain relief after laparotomy. Br J Surg. 2001 Mar;88(3):357-9. doi: 10.1046/j.1365-2168.2001.01717.x. PMID 11260098
- [Background] Clinical Outcomes of Surgical Therapy Study Group; Nelson H, Sargent DJ, Wieand HS, Fleshman J, Anvari M, Stryker SJ, Beart RW Jr, Hellinger M, Flanagan R Jr, Peters W, Ota D. A comparison of laparoscopically assisted and open colectomy for colon cancer. N Engl J Med. 2004 May 13;350(20):2050-9. doi: 10.1056/NEJMoa032651. PMID 15141043
- [Background] Ashcraft EE, Baillie GM, Shafizadeh SF, McEvoy JR, Mohamed HK, Lin A, Baliga PK, Rogers J, Rajagopalan PR, Chavin KD. Further improvements in laparoscopic donor nephrectomy: decreased pain and accelerated recovery. Clin Transplant. 2001;15 Suppl 6:59-61. doi: 10.1034/j.1399-0012.2001.00011.x. PMID 11903389
- [Background] Melzack R. The McGill Pain Questionnaire: major properties and scoring methods. Pain. 1975 Sep;1(3):277-299. doi: 10.1016/0304-3959(75)90044-5. PMID 1235985